CLINICAL TRIAL: NCT01776489
Title: The Role of Sphingosine-1-phosphate in Food Allergy - Biomarker for Disease Severity and Anaphylaxis Outcome
Brief Title: Evaluation of the Sphingolipid Metabolite S1P as a Novel Biomarker in Food Allergy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Eva Untersmayr-Elsenhuber, Assoc. Prof., Dr., Medical University of Vienna
Other Study IDs: 119/2011; KLI 284-B00 (Other Grant/Funding Number: Austria Science Fund)
Record Dates: First submitted 2013-01-21; First posted 2013-01-28 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Food Allergy; Anaphylaxis
Keywords: Food allergy; Sphingosine-1-phosphate; Biomarker; Double-blind placebo-controlled food challenge; Anaphylaxis
MeSH Terms: conditions — Food Hypersensitivity; Anaphylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- food allergic: positive reaction during DBPCFC
- Non-food allergic: no reaction during DBPCFC

SUMMARY:
Food allergies represent an increasing health concern in the industrialized countries and especially affect pediatric patients. In this population adverse reactions against food compounds can lead to anaphylactic reactions. Despite substantial research efforts, clinical markers predicting disease severity and symptoms are missing to date.

Recent studies have revealed that sphingolipids, especially sphingosine-1-phosphate (S1P), play an essential role in allergy. It was reported that asthmatic patients have higher S1P levels in bronchiallavage fluids after allergen challenge. First experimental studies revealed a correlation of S1P and the outcome of anaphylaxis. Furthermore, we have shown in our recent mouse study that S1P homeostasis is pivotal for food allergy induction and effector cell response. Therefore, it is the aim of the presented pilot project to evaluate whether S1P serum titers are altered in food allergic children and if the S1P levels correlate with the outcome of anaphylaxis during double blind placebo controlled food challenges (DBPCFCs).

ELIGIBILITY:
Inclusion Criteria:

* Patients between 1-17 years who have been reported to suffer from food allergic reactions and who are subjected to DBPCFC or open provocation
* Patients who are diagnosed by elevated allergen specific IgE and/or positive skin prick testing
* Willingness to participate in the study

Exclusion Criteria:

* Refusal to participate in the study
* Non-IgE-mediated food allergy

Ages: 12 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children (age 1-17 years) being in medical care at the allergy clinic of the Department of Pediatrics and Adolescent Medicine of the Medical University of Vienna for food related immediate type symptoms (nausea, abdominal pain, vomiting, diarrhea or local symptoms like burning, swelling, itching and erythema) immediately after ingestion of food compounds will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2011-12; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
S1P in allergic and non-allergic patients before and after challenge | up to 3 years
  The primary endpoint of this study is the measurement of S1P in allergic and non-allergic patients before and after challenge.

SECONDARY OUTCOMES:
Evaluation of allergic mediators and correlation with S1P levels | up to 3 years
  Evaluation of allergic mediators like histamine, human mast cell tryptase and eosinophil cationic protein and correlate these results with the levels of S1P within the group and between allergic and non-allergic patients

CONTACTS AND LOCATIONS:
Overall Officials: Eva Untersmayr-Elsenhuber, MD, PhD, Principal Investigator — Medical University Vienna, Department of Pathophysiology and Allergy Research
Locations (1):
- Medical University Vienna, Department of Pediatrics and Adolescent Medicine, Vienna, Austria

REFERENCES:
- [Background] Diesner SC, Olivera A, Dillahunt S, Schultz C, Watzlawek T, Forster-Waldl E, Pollak A, Jensen-Jarolim E, Untersmayr E, Rivera J. Sphingosine-kinase 1 and 2 contribute to oral sensitization and effector phase in a mouse model of food allergy. Immunol Lett. 2012 Jan 30;141(2):210-9. doi: 10.1016/j.imlet.2011.10.006. Epub 2011 Oct 14. PMID 22020265
- [Background] Olivera A, Eisner C, Kitamura Y, Dillahunt S, Allende L, Tuymetova G, Watford W, Meylan F, Diesner SC, Li L, Schnermann J, Proia RL, Rivera J. Sphingosine kinase 1 and sphingosine-1-phosphate receptor 2 are vital to recovery from anaphylactic shock in mice. J Clin Invest. 2010 May;120(5):1429-40. doi: 10.1172/JCI40659. Epub 2010 Apr 19. PMID 20407207
- [Background] Olivera A, Mizugishi K, Tikhonova A, Ciaccia L, Odom S, Proia RL, Rivera J. The sphingosine kinase-sphingosine-1-phosphate axis is a determinant of mast cell function and anaphylaxis. Immunity. 2007 Mar;26(3):287-97. doi: 10.1016/j.immuni.2007.02.008. Epub 2007 Mar 8. PMID 17346996
- [Background] Ammit AJ, Hastie AT, Edsall LC, Hoffman RK, Amrani Y, Krymskaya VP, Kane SA, Peters SP, Penn RB, Spiegel S, Panettieri RA Jr. Sphingosine 1-phosphate modulates human airway smooth muscle cell functions that promote inflammation and airway remodeling in asthma. FASEB J. 2001 May;15(7):1212-4. doi: 10.1096/fj.00-0742fje. No abstract available. PMID 11344091
- See also: study center — http://www.meduniwien.ac.at/ipa
- See also: study center — http://www.meduniwien.ac.at/kinderklinik/
- See also: project homepage — http://www.gastrointestinal.at